CLINICAL TRIAL: NCT03047057
Title: Effect of Lidocaine Infusion on Acute Rehabilitation After Radical Cystectomy
Brief Title: Lidocaine Infusion in Radical Cystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM12017
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): IV Lidocaine infusion
  Interventions: Drug: Lidocaine
- Control (Placebo Comparator): IV normal saline infusion
  Interventions: Drug: IV normal saline

INTERVENTIONS:
Drug: Lidocaine — IV Lidocaine infusion
  Arms: Lidocaine
Drug: IV normal saline — IV normal saline infusion
  Other Names: normal saline
  Arms: Control

SUMMARY:
Radical cystectomy (RC) remains the gold standard for treatment of patients with muscle invasive bladder cancer, or recurrent high grade non-muscle invasive bladder cancer. Nowadays, enhanced recovery pathway is used to decrease morbidity and improve acute rehabilitation after RC. Postoperative ileus is the most frequent reason for prolonged hospital stay following cystectomy.

DETAILED DESCRIPTION:
Radical cystectomy remains the gold standard for treatment of patients with muscle invasive bladder cancer, or recurrent high grade non-muscle invasive bladder cancer. The high rates of morbidity and mortality reflect the fact that the majority of patients undergoing this procedure are elderly patients with multiple comorbidities. Postoperative ileus is the most frequent reason for prolonged hospital stay following cystectomy. To reduce the risk of ileus, prokinetics such as metoclopramide should be used postoperatively. Local anesthetics exert their actions as local anesthesia and antiarrhythmic through Na channels blocking but still have many other important actions through other receptors (e.g., m1 muscarinic receptors) that occur at very low plasma levels compared to levels needed for Na channels blocking, one of these actions is the anti-inflammatory effect against surgical stress response. Several randomized studies found that i.v. lidocaine shortens duration of postoperative ileus and some of it reported decreased postoperative pain with i.v. lidocaine, so they recommended i.v. lidocaine as a safe, simple, and less invasive method for management of postoperative ileus and equal to postoperative epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 yr ASA class I,II, and III Elective radical cystectomy

Exclusion Criteria:

* Allergy to the study medication, pre-existing chronic pain at any site requiring treatment, Psychiatric disease, hepatic or renal impairment, seizure disorder requiring medication within the previous 2 years

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Postoperative return of gastrointestinal (GI) function | 15 day
  Time to the first defecation

SECONDARY OUTCOMES:
Postoperative Pain | 72 hours after surgery
  a 10 cm visual analog pain scale (VAS) at rest and during mobilization

CONTACTS AND LOCATIONS:
Locations (1):
- Seham Mohamed Moeen Ibrahim, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moeen SM, Moeen AM. Usage of Intravenous Lidocaine Infusion with Enhanced Recovery Pathway in Patients Scheduled for Open Radical Cystectomy: A Randomized Trial. Pain Physician. 2019 Mar;22(2):E71-E80. PMID 30921979